CLINICAL TRIAL: NCT06342063
Title: The Effects of Preoperative Blood Flow Restriction Training in Patients Undergoing ACL Reconstruction: A Pilot Randomized Control Trial
Brief Title: The Effects of Preoperative Blood Flow Restriction Training in Patients Undergoing ACL Reconstruction
Acronym: BFRACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0070-E
Record Dates: First submitted 2024-03-11; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: ACL Injury; Sports Physical Therapy
Keywords: Blood Flow Restriction; Preconditioning; Rehab; ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Patients were recruited and randomized to one of the two treatment arms.
Who Masked: Outcomes Assessor
Masking Description: Outcome measurement was blinded to participant intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy with Blood Flow Restriction Group (Active Comparator): This group underwent a physiotherapy protocol while using Blood Flow Restriction adjunctive therapy prior to ACL reconstruction.
  Interventions: Device: Blood Flow Restriction Therapy
- Physiotherapy without Blood Flow Restriction Group (Sham Comparator): This group underwent a physiotherapy protocol without using Blood Flow Restriction adjunctive therapy prior to ACL reconstruction.
  Interventions: Device: Blood Flow Restriction Therapy Sham

INTERVENTIONS:
Device: Blood Flow Restriction Therapy — Patients wear a personalized tourniquet pressure system on their involved thigh while they perform a series of leg press machine exercises. This tourniquet is inflated.
  Other Names: BFR
  Arms: Physiotherapy with Blood Flow Restriction Group
Device: Blood Flow Restriction Therapy Sham — Patients wear a personalized tourniquet pressure system on their involved thigh while they perform a series of leg press machine exercises. This tourniquet is not inflated.
  Other Names: Sham BFR Comparison Group
  Arms: Physiotherapy without Blood Flow Restriction Group

SUMMARY:
This prospective feasibility study is designed to assess pre-operative BFR in patients awaiting ACL reconstruction. This study will serve the following: (1) to determine if BFR improves strength testing prior to surgery and (2) to determine if BFR reduces QF muscle group atrophy prior to surgery. Additionally, preliminary results on pre-operative clinical and quality of life scores will be collected. If this study shows encouraging results, it will serve as a template for a more comprehensive randomized control trial.

DETAILED DESCRIPTION:
Quadriceps femoris (QF) muscle function is an integral factor in the rehabilitation and overall outcome after lower extremity injury or surgical intervention. Atrophy of this muscle group is a common finding in patients undergoing anterior cruciate ligament (ACL) reconstruction. This is due to the immobility prior to surgery, vascular ischemia caused by a tourniquet intra-operatively and inability to perform high load strength training in the early post-operative period. A deficit in QF muscle strength can result in excessive joint loading and be a contributing factor in the early onset of osteoarthritis of the knee. It should be noted that a loss of strength in this primary knee extensor mechanism muscle group can persist for up to 2 years after surgery. Thus, the reduction of QF atrophy and maintenance of strength during an intervention such as an ACL reconstruction has large implications for the overall post-operative outcome and natural history of the knee joint.

In order to combat the challenges of muscle atrophy for patients with an ACL injury, blood flow restriction (BFR) training has been shown to have beneficial effects in the post-operative period specifically. The process of using BFR therapy involves the application of an extremity tourniquet to occlude venous outflow and restrict arterial inflow. Thus, an anaerobic environment is created to promote muscle hypertrophy by having cells upregulate cell signalling, protein synthesis and ultimately myogenic proliferation. The use of BFR during lower extremity rehabilitation has shown that its simultaneous use with low load resistance training can have similar hypertrophic effects to isolated high load resistance training. This is ideal for patients who are initially unable to perform high intensity exercises shortly after an ACL reconstruction surgery, but are attempting to reduce overall QF atrophy.

However, the use of BFR in the pre-operative period has yet to be well established. Preconditioning with an ischemic environment may provide an effective way to reduce QF atrophy with low load exercises while awaiting surgery. Additionally, having a period of sensitization with anaerobic conditions prior to surgery, may provide some resistance to the damaging effects of a tourniquet intra-operatively. The limited studies that have attempted to use BFR therapy prior to ACL surgery have had short intervention periods, small sample sizes and outcome variables that have not assessed overall clinical outcome. If BFR in the pre-operative setting can be shown to provide beneficial effects, it will be a valuable tool in maximizing the overall outcome of patients undergoing ACL reconstruction.

This prospective feasibility study has been designed to assess pre-operative BFR in patients awaiting ACL reconstruction. This study will serve the following: (1) to determine if BFR improves strength testing prior to surgery and (2) to determine if BFR reduces QF muscle group atrophy prior to surgery. Additionally, preliminary results on pre-operative clinical and quality of life scores will be collected. If this study shows encouraging results, it will serve as a template for a more comprehensive randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Sagittal Knee instability caused by ACL tear requiring surgical reconstruction
* Minimum 4 weeks since the time of injury
* Age 18 to 50 years

  * Range of motion required

    ▪ Active extension deficit <5o, Active flexion > 120o
  * No previous surgery to affected knee

Exclusion Criteria:

* Functional impairment (neuro disease, gait abnormality, ambulatory aids at baseline)
* Severe spine or lower limb injuries
* Comorbidities including cardiovascular, respiratory or metabolic disease, blood coagulation disorders, current smoker

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Biodex Strength Testing | Baseline testing 1 day prior to physiotherapy initiation and Post intervention testing performed 1 day after physiotherapy completion but before ACL surgery.
  Quadriceps and Hamstring Muscle Strength and Endurance testing. Maximal peak torque (FT-LBS) was recorded for both knee flexion and extension at 60 degrees / second (indicative of strength) and 180 degrees / second (indicative of endurance).

SECONDARY OUTCOMES:
Short Form Health Survey 12 (SF-12) | Baseline testing 1 day prior to physiotherapy initiation and Post intervention testing performed 1 day after physiotherapy completion but before ACL surgery.
  Patient Reported Outcome Measure. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline testing 1 day prior to physiotherapy initiation and Post intervention testing performed 1 day after physiotherapy completion but before ACL surgery.
  Patient Reported Outcome Measure. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.

CONTACTS AND LOCATIONS:
Overall Officials: John Theodoropoulos, MD, FRCSC, Principal Investigator — Dovigi Sports Medicine Clinic, Mount Sinai Hospital, Toronto, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wengle L, Migliorini F, Leroux T, Chahal J, Theodoropoulos J, Betsch M. The Effects of Blood Flow Restriction in Patients Undergoing Knee Surgery: A Systematic Review and Meta-analysis. Am J Sports Med. 2022 Aug;50(10):2824-2833. doi: 10.1177/03635465211027296. Epub 2021 Aug 18. PMID 34406084

DOCUMENTS (2):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT06342063/Prot_000.pdf
  • Informed Consent Form (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT06342063/ICF_001.pdf